CLINICAL TRIAL: NCT04506632
Title: COST-NHS: COvid Burden in STaff Working in the NHS: A Study to Assess the Mental Health Burden of the COVID-19 Pandemic on NHS Healthcare Staff
Brief Title: Burden for STaff Working in the NHS
Acronym: COST-NHS
Status: Active, not recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH21373
Record Dates: First submitted 2020-07-21; First posted 2020-08-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Mental Health Burden
Keywords: COVID-19; Coronavirus; NHS staff; Mental health
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The COVID-19 crisis began in China in December 2019 and was declared a pandemic by the World Health Organisation on March 11th 2020. The pandemic has changed the way that clinicians interact with and treat patients overnight. Staff within the NHS will be under high levels of stress due to the increased needs and worse outcomes of work as they are shielding or self-isolating and may feel helpless and guilty. The psychological impact of the pandemic will be prolonged and varied. It is vital that Investigators increase understanding as much as possible to support NHS staff.

The aim of this survey is to examine the possible mental health burden on NHS staff as a result of the COVID-19 pandemic and how these change as the pandemic progresses. By understanding these effects, it will allow researchers to identify recommendations to allow support mechanisms to be put in place for NHS staff, to better manage this and future pandemics and similar crises.

Investigators are aiming to sample several cohorts of NHS staff including a subset of staff who are shielding. Staff will be asked to complete a series of online surveys at multiple timepoint: on study initiation, 1 month later and then 3 months after the pandemic has ceased in the UK. Additional timepoints may be added depending on the length and severity of the pandemic.

The main outcomes will be tracking changes in mental health measurements at the pre-defined timepoints. This work will allow Investigators to produce recommendations about the increased mental health support that NHS staff will need. If a need is demonstrated then an interventional research project will be designed and implemented.

DETAILED DESCRIPTION:
The aim of this survey is to examine the possible mental health burden on NHS staff as a results of the coronavirus COVID-19 pandemic and how these change as the pandemic progresses. By understanding these effects, it will allow Investigators to identify recommendations to allow appropriate support mechanisms to be put in place for NHS staff, to better manage this and future pandemics and similar crises.

Method:

Investigators aim to sample several cohorts of staff across the NHS. A subset of participants will include NHS staff that are currently shielding - they are self-isolating due to being identified as part of the at-risk/vulnerable members of society. The aim will be to survey a minimum of 100 members of staff. Introductory emails will be sent out to NHS staff using the hospital email system. Potential participants will be asked to read a participant information sheet and provide informed consent to participate in the subsequent survey.

Staff within the NHS will be asked to complete a series of surveys at multiple timepoints. The survey link will be circulated to staff with the introductory email. It will be sent at the following time points with a reminder to all on each occasion after 5 days: on study initiation, 1 month later and then 3 months after the pandemic has ceased in the UK. Additional timepoints may be added depending on the length and severity of the pandemic.

Qualtrics software will be used to host and administer the survey. The variables to be measured are:

Demographics (At first survey only): Age, sex, ethnic status, socio-economical status, religious identification and occupation.

Exposure to COVID-19 Mental health: The investigators will assess depression with 9 items (PHQ-9); anxiety with 7 items (GAD-7); paranoia (short Green paranoia scale), traumatic stress, somatic symptoms (PHQ-15); conspiracy mentality and social interactions (The loneliness scale).

Mediating psychological variables: Locus of control, death anxiety, 10 item Cognitive Reflection Task of analytical reasoning and personality traits 9 Big-five short version.

The surveys should take approximately 10 minutes to complete. Participants will be informed that should they feel distressed by the questions raised in the survey, that they should seek support from the providers in the introductory email. Participants will be able to withdraw from the study and any timepoint without providing a reason.

The participants anonymised data will be analysed by Professor Bentall's team at the University of Sheffield and stored on a secure, University server. The main outcomes of the study will be tracking changes in mental health measurements at the pre-defined timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 16 years or over
* Participants must be working in the NHS
* NHS staff that are shielding will be eligible to participate
* NHS staff that are self-isolating will be eligible to participate
* Able and willing to provide informed consent
* Able to read and understand English

Exclusion Criteria:

• Participants will not be excluded on any other basis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit NHS staff that are working during the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Depression | UP to 3 months after the pandemic ends in the UK
  We will assess depression with 9 items (PHQ-9);
Changes in Anxiety | UP to 3 months after the pandemic ends in the UK
  measured by GAD-7
Changes in feelings of paranoia | UP to 3 months after the pandemic ends in the UK
  measured by the short Green paranoia scale
Traumatic Stress | UP to 3 months after the pandemic ends in the UK
  As measured by PHQ-15
conspiracy mentality and social interactions | UP to 3 months after the pandemic ends in the UK
  as measured by the loneliness scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Danson, Professor, Study Director — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No